CLINICAL TRIAL: NCT03943173
Title: NOW: Neoadjuvant Olaparib Window Trial in Newly Diagnosed BRCA-Mutant Ovarian Cancer
Brief Title: Olaparib in Treating Patients With Newly Diagnosed BRCA-Mutant Ovarian, Primary Peritoneal, or Fallopian Cancer Before Surgery
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0775; NCI-2019-00503 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0775 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-21; First posted 2019-05-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: BRCA-Mutated Ovarian Carcinoma; BRCA1 Gene Mutation; BRCA2 Gene Mutation; High Grade Fallopian Tube Serous Adenocarcinoma; High Grade Ovarian Serous Adenocarcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Stage III Fallopian Tube Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage IIIA Fallopian Tube Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Primary Peritoneal Cancer AJCC v8; Stage IIIA1 Fallopian Tube Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Fallopian Tube Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Fallopian Tube Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Primary Peritoneal Cancer AJCC v8; Stage IIIC Fallopian Tube Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Drug Therapy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. After treatment, patients either undergo surgery then receive standard chemotherapy for up to 4 cycles or receive standard chemotherapy within 14 days for up to 4 cycles then undergo surgery in the absence of disease progression or unacceptable toxicity at the discretion of the treating physician.
  Interventions: Drug: Chemotherapy; Drug: Olaparib; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Chemotherapy — Given standard chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Drug: Olaparib — Given PO
  Other Names: AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This early phase I trial studies how well olaparib works in treating patients with newly diagnosed BRCA-mutant ovarian, primary peritoneal, or fallopian cancer before surgery. Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of daily olaparib given in the neoadjuvant setting in women with primary advanced high grade non-mucinous epithelial ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. Estimate efficacy of olaparib given in the neoadjuvant setting using response rate (by Response Evaluation Criteria in Solid Tumors [RECIST] in subjects with measurable disease).

II. Estimate proportion of subjects able to proceed immediately to interval tumor reductive surgery (without chemotherapy).

III. Determine progression-free survival (PFS). IV. Determine complete pathologic response rate at the time of surgery. V. Determine the toxicity of daily olaparib given in the neoadjuvant setting. VI. Evaluate the toxicity of chemotherapy given after neoadjuvant olaparib. VII. Measure longitudinal symptom burden of study subjects treated with neoadjuvant olaparib and chemotherapy after olaparib.

EXPLORATORY OBJECTIVES:

I. Explore deoxyribonucleic acid (DNA) copy number and level of ribonucleic acid (RNA) and protein expression in homologous recombination-related pathways before and after treatment with olaparib in women with primary advanced high grade non-mucinous epithelial ovarian, fallopian tube, or primary peritoneal cancer.

II. Correlate molecular results to clinical endpoints including response and survival.

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. After treatment, patients either undergo surgery then receive standard chemotherapy for up to 4 cycles or receive standard chemotherapy within 14 days for up to 4 cycles then undergo surgery in the absence of disease progression or unacceptable toxicity at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the United States of America [USA]) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Histology showing high-grade epithelial non-mucinous ovarian, primary peritoneal, or fallopian tube cancer
* Documented BRCA pathway mutations
* No prior treatment for primary advanced (stage III or IV) epithelial ovarian, primary peritoneal, or fallopian tube carcinoma such as irradiation, chemotherapy, hormonal therapy, immunotherapy, investigational therapy, surgery, and/or other concurrent agents or therapies
* A disposition to neoadjuvant chemotherapy (NACT) with planned interval tumor reductive surgery after 3 complete cycles of treatment
* Have measurable disease based on RECIST version 1.1 or evaluable disease. Measurable disease is defined at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each "target" lesion must be > 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or > 10 mm when measured by spiral CT. Evaluable disease includes nonmeasurable lesions, ascites, pleural effusion
* Peripheral neuropathy grade 0 or 1 by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >= 16 weeks
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as: amenorrheic for 1 year or more following cessation of exogenous hormonal treatments, luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50, radiation-induced oophorectomy with last menses > 1 year ago, chemotherapy-induced menopause with > 1 year interval since last menses, or surgical sterilization (bilateral oophorectomy or hysterectomy). Women of childbearing potential (WoCBP) must utilize acceptable contraception for two weeks before the first dose of olaparib, for the duration of the study, and for at least 6 months after the last dose of olaparib
* Hemoglobin >= 10.0 g/dL (with no blood transfusion in the past 28 days) (measured within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 109/L (> 1500 per mm3) (measured within 28 days prior to administration of study treatment)
* Platelet count >= 100 x 109/L (> 100,000 per mm3) (measured within 28 days prior to administration of study treatment)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) (measured within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN unless liver metastases are present, in which case it must be =< 5 x ULN (measured within 28 days prior to administration of study treatment)
* Serum creatinine clearance (CrCL) >= 51 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of CrCL (measured within 28 days prior to administration of study treatment)

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrollment in the present study
* Prior treatment for ovarian, fallopian tube, or primary peritoneal cancer
* Histology showing mucinous or low grade epithelial carcinoma
* Participation in another clinical study with an investigational product (IP) during the last 4 weeks
* History of another primary malignancy except for: malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, and/or adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, mean QT interval corrected for heart rate with Fridericia's correction (QTcF) prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Any unresolved toxicity (> CTCAE grade 2) from previous anti-cancer therapy, excluding alopecia
* History of hypersensitivity to olaparib or its excipients
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV) or otherwise immunocompromised subjects, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* History of leptomeningeal carcinomatosis
* Subjects who are pregnant and/or breast-feeding
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of subject safety or study results
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids. The subject can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Subjects with uncontrolled seizures
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML)
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Any previous treatment with PARP inhibitor, including olaparib
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort ) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable outside of 28 days prior to treatment)
* Non-English speakers will be excluded from participating in the patient-reported outcomes component of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Feasibility of olaparib | Up to 1 year
  Feasibility defined by number of subjects who are able to receive two cycles of PARP inhibition without unacceptable toxicity or disease progression (new disease or increase of CA125 from baseline > 50%). Will be analyzed using descriptive statistics. Will be estimated using a 90% credible interval

SECONDARY OUTCOMES:
Response rate | U to 1 year
  For categorical endpoints, standard descriptive statistics, including frequency table and exact 95% confidence intervals will be computed using the Clopper-Pearson method.
Complete pathologic response | For up to 1 year
  For categorical endpoints, standard descriptive statistics, including frequency table and exact 95% confidence intervals will be computed using the Clopper-Pearson method.
Incidence of adverse events | For up to 1 year
  For categorical endpoints, standard descriptive statistics, including frequency table and exact 95% confidence intervals will be computed using the Clopper-Pearson method.
Symptom burden and health status | For up to 1 year
  Will be assessed by the MD Anderson Symptom Inventory (MDASI) ."For categorical endpoints, standard descriptive statistics, including frequency table and exact 95% confidence intervals will be computed using the Clopper-Pearson method.
Progression-free survival | Up to 1 year
  Summarized using descriptive statistics, including Kaplan-Meier curve and estimates.
Symptom burden and health status | For up to 1 year
  Will be assessed by EuroQol 5-dimension. For categorical endpoints, standard descriptive statistics, including frequency table and exact 95% confidence intervals will be computed using the Clopper-Pearson method.
Symptom burden and health status | For up to 1 year
  Will be assessed by 5-level (EQ-5D-5L) instruments. For categorical endpoints, standard descriptive statistics, including frequency table and exact 95% confidence intervals will be computed using the Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pending discussions with AstraZeneca regarding the level and quantity of data that may be shared. Discussions will also include potential modifications of the contract to allow for data sharing.

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org